CLINICAL TRIAL: NCT05442970
Title: An Epidemiologic, Prospective, Single Center Cohort Study for the Improvement of Atrial Fibrillation Risk Stratification in High Risk Individuals
Brief Title: Cohort Study for Atrial Fibrillation Risk Stratification
Acronym: AFHRI
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: AFHRI
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sophisticated biobank including DNA, RNA, cells, and serum/plasma for comprehensive genetic, gene expression and proteomic studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AFHRI is planned as a prospective, single-center cohort study in patients at high risk of AF.

DETAILED DESCRIPTION:
The primary aim of the study is to evaluate and improve atrial fibrillation risk prediction, which takes into account clinical, psycho-social, environmental and lifestyle-risk factors, protein patterns and genetic variability in addition to the classical risk factors with respect to the primary endpoint, AF (paroxysmal or permanent).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years;
* Personally signed informed consent

Exclusion Criteria:

* Insufficient knowledge of the German language, in order to understand study documents and computer assisted interview without translation;
* Physical or psychological incapability to cooperate in the investigations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 1/1 selection
Study Population: Outpatient cardiology sample at risk for AF. Recruitment in a single center design, at the Department of Cardiology, University Medical Center Hamburg-Eppendorf.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Incident atrial fibrillation | up to 4 years
  12-lead Electrocardiogram (ECG) tracing, diagnosis of AF will be made if at least two cardiologists verify the rhythm abnormality using clinic visit, outside physician or hospital records, or ambulatory ECG reports.

SECONDARY OUTCOMES:
Myocardial infarction | up to 4 years
  Typical rise and gradual fall (Troponin) or more rapid rise and fall (CK-MB) of biochemical markers of myocardial necrosis
Cardiovascular death | up to 4 years
  if no other underlying cause of death is diagnosed: hypertension, coronary heart disease, other cardiovascular disease, atherosclerosis, diabetes mellitus, dyslipidemia, obesity, sudden death and cardiac symptoms
Heart failure | up to 4 years
  echocardiography including Doppler-flow measurement

CONTACTS AND LOCATIONS:
Overall Officials: Renate B Schnabel, Prof., Principal Investigator — Department of Cardiology, University Medical Center Hamburg-Eppendorf
Locations (1):
- Department of Cardiology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Owing to propriety nature, supporting data cannot be made available openly. Further information about the data and access conditions is available uppon request

REFERENCES:
- [Result] Assum I, Krause J, Scheinhardt MO, Muller C, Hammer E, Borschel CS, Volker U, Conradi L, Geelhoed B, Zeller T, Schnabel RB, Heinig M. Tissue-specific multi-omics analysis of atrial fibrillation. Nat Commun. 2022 Jan 21;13(1):441. doi: 10.1038/s41467-022-27953-1. PMID 35064145